CLINICAL TRIAL: NCT02502292
Title: Sustainable Health Systems Through Health Literacy for Healthy Aging
Brief Title: Innovative Policies for Healthy Aging
Acronym: IROHLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacobs University Bremen gGmbH (Other)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Sonia Lippke, Professor of Health Psychology, Jacobs University Bremen gGmbH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FP7/2007-2013
Record Dates: First submitted 2015-07-06; First posted 2015-07-20 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Health Behavior; Attitude to Health; Impaired Health
Keywords: Health Literacy; Health Ageing; Health Literacy Interventions; IROHLA; Photo Novel Study
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention: Fotonovela (Experimental): The Photo Novel Intervention is presented to users of four different facilities (sports clubs, senior homes) who are older than 50 years. The researchers welcome scheduled eligible participants, introduce the study and ask them for their consent. Afterwards, the participants are asked to fill in the questionnaire. Then, participants are randomized to one of the four groups and are presented with the photo novel or traditional brochure either as a hard copy brochure or as pdf on a tablet computer (2x2 group design). They are instructed to read the material in their own pace and answer the accompanying questions after each story / tip.and the accompanying questionnaire.
  Interventions: Behavioral: Fotonovela

INTERVENTIONS:
Behavioral: Fotonovela — Comparing fotonovela brochure to traditional brochure, as a template communicative behaviors embedded in a picture story where the older people could use before and during primary care consultations with their GP. Relevant communicative behaviors will include 'asking questions', 'expressing lack of or misunderstanding', 'expressing uncertainty', 'expressing preferences and needs' and other relevant communicative behaviors which are based on communication theory / literature and on the output of the focus group discussions.
  The researchers will randomly assigned the participants into four groups as described earlier. Mainly to identify the outcomes of the comparison between fotonovela and traditional brochure in both traditional hard-copy and in tablet.

SUMMARY:
In this study, the investigators evaluate an intervention aiming to increase participation and communication of older adults during primary care consultations with their General Practitioner(GP). The investigators are particularly interested in a Photo novel tool with this aim. Photo novels are picture stories, which have the advantage of using a familiar narrative format, thereby possibly increasing comprehension, personal involvement and motivation and self-efficacy to perform the relevant behaviors by offering role models (story characters that are similar to older adults themselves). The patient perspective on doctor-patient communication is underrepresented in most research. This study aims to incorporate the patient perspective in different ways: in addressing their needs and barriers during focus group discussions, in collecting their communication strategies and solutions to these barriers in the role play exercise, in involving them in developing the photo novel, and in studying their responses to the photo novel in the evaluation study the investigators describe in this research proposal.

DETAILED DESCRIPTION:
In this study, the researchers evaluate an intervention aiming to increase participation and communication of older adults during primary care consultations with their General Practitioner (GP). The researchers are particularly interested in a Photo novel tool with this aim. Photo novels are picture stories, which have the advantage of using a familiar narrative format, thereby possibly increasing comprehension, personal involvement and motivation and self-efficacy to perform the relevant behaviors by offering role models (story characters that are similar to older adults themselves). The patient perspective on doctor-patient communication is underrepresented in most research. This study aims to incorporate the patient perspective in different ways: in addressing their needs and barriers during focus group discussions, in collecting their communication strategies and solutions to these barriers in the role play exercise, in involving them in developing the photo novel, and in studying their responses to the photo novel in the evaluation study the researchers describe in this research protocol.

Aim of the intervention (the Photo novel) is to:

1. increase older adults' awareness of their needs and barriers in conversations with their GP;
2. improve older adults' access to information by enabling them to ask different and more questions to their GP;
3. increase older adults' problem solving abilities during conversations with their GP to ensure better self-management of health issues.
4. find out which format is most efficacious

This could include being honest about limited understanding, asking for more information to enable or improve shared decision making during consultation or to enable or improve self-management after consultation. This could also include filtering information and enabling patients to determine relevance of information. Furthermore, this could include strategies to translate advice into concrete actions, e.g. transforming 'knowing that' into 'knowing how' (I know / understand that I have to use less salt but… How to… decrease salt-intake in daily life?) In our photo novel, the researchers will provide older adults with 'template communicative behaviors' embedded in a picture story they can use before and during primary care consultations with their GP. Relevant communicative behaviors will include 'asking questions', 'expressing lack of or misunderstanding', 'expressing uncertainty', 'expressing preferences and needs' and other relevant communicative behaviors that will be identified during the focus group discussions with older adults and their informal care givers. These relevant communicative behaviors are embedded within different relevant domains, based on communication theory / literature and on the output of the focus group discussions. The seven scenarios are linked to the endpoints of medical communication framework developed by Haes and Bensing.

The researchers propose to evaluate the effectiveness of the photo novel using an Experimental Design, including both quantitative and qualitative measurements. This combination of measurements will provide us with insight with regard to three important Research Questions:

1. To what extent is a photo novel an effective tool / intervention to empower older adults in their conversations with their GP compared to a traditional brochure containing tips on GP-patient communication?
2. Which elements or domains included in the photo novel are effective and why?
3. Which narrative / theoretical mechanisms account for the effectiveness of the photo novel ?

The researchers will recruit older adult participants (>50 years), who live in areas indicative of limited or marginal health literacy. The researchers perform the following procedure for recruitment. The researchers recommend to build relationships with GP practices, healthcare organizations and community organizations and ask them for their cooperation during a pre-established period of time. The researchers pay careful attention to this part of our study, e.g. carefully design recruitment wording: 'We are conducting a study to improve the relationship/ conversations with your GP, as a way to make sure the health care you receive is improved. We invite you to participate in this study. Would you like to participate?' Participants will be asked to come to a neutral setting, for example within the University, or will be visited in a community building, to take part in our study. Based on their consent to participate, a schedule is developed with eligible patients. Participants will be randomized to one of the two conditions and will be presented with the photo novel or traditional brochure either presented as a hard copy brochure or as pdf on a tablet computer (2x2 factorial design) and the accompanying questionnaire. The researchers aim for participants of different ages.

ELIGIBILITY:
Inclusion Criteria:

* Areas indicative of limited or marginal health literacy
* Carry out in a neutral setting

Exclusion Criteria:

* Eye-sight or hearing disabled people. This is because this study requires participants have the ability to read and watch and listen to videos.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Health literacy will be assessed by questions in a questionnaire | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Lippke, Prof.Dr., Principal Investigator — Jacobs University Bremen; Ruth Koops van 't Jagt, Msc., Principal Investigator — Reichuniversität Groningen/UMCG
Locations (1):
- Jacobs University Bremen gGmbH, Bremen, Germany

REFERENCES:
- [Derived] Tan SL, Whittal A, Lippke S. Testing a Photo Story Intervention in Paper Versus Electronic Tablet Format Compared to a Traditional Brochure Among Older Adults in Germany: Randomized Controlled Trial. JMIR Aging. 2018 Dec 6;1(2):e12145. doi: 10.2196/12145. PMID 31518254
- See also: Homepage of the official website — http://www.irohla.eu/